CLINICAL TRIAL: NCT00860210
Title: Pilot Feasibility Study of the Neurostep™ System in Subjects With Gait Disorder Secondary to CNS Lesion.
Brief Title: Pilot Study Assessing the Feasibility of Treating Foot Drop With the Neurostep™ System.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurostream Technologies G.P. (Industry)
Responsible Party: Neurostream Technologies, G.P., Neurostream Technologies, G.P.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VHB-PFS-NSS III; VHB-PFS-NSS III-SS01-PRT; VHB-PFS-NSS III-SS02-PRT; VHB-PFS-NSS III-SS03-PRT; VHB-PFS-NSS III-SS04-PRT
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2010-04-12 (Estimated); Status verified 2010-04

CONDITIONS: Stroke; Craniocerebral Trauma
MeSH Terms: conditions — Stroke; Craniocerebral Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Neurostep™ System — The Neurostep™ System is a neurostimulation investigational medical device. The entire system is designed to be implanted into the subject's leg via a surgical procedure, during which electrodes are attached to the peripheral nerves responsible for sensing and stimulating the proper muscles that lift the foot during normal walking.
  Other Names: Neurostep

SUMMARY:
This pilot feasibility study is assessing the safety and technical performance of the Neurostep™ System for the restoration of independent gait in subjects with gait disorder (i.e. foot drop) secondary to a CNS lesion (e.g. stroke).

DETAILED DESCRIPTION:
The Neurostep™ System is a neurostimulation investigational medical device. The entire system is designed to be implanted into the subject's leg via a surgical procedure, during which electrodes are attached to the peripheral nerves responsible for sensing and stimulating the proper muscles that lift the foot during normal walking.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a unilateral gait disorder as a result of a specified CNS lesion (e.g., stroke)with stable neurological deficit for at least 6 months
* Medically stable, able to and agree to undergo a surgery
* Able to stand and walk at least 5 meters
* Agree to attend frequent study scheduled visits
* Able to provide verbal or written feedback
* Have provided written informed consent
* Have intact tibial and common peroneal nerves

Exclusion Criteria:

* Pregnant or nursing women
* Medically insufficiently stable to undergo surgery
* Poor range of motion of affected ankle or fixed ankle
* Foreseen need for Magnetic Resonance Imaging (MRI)
* Significant mental or psychiatric impairment
* Cannot understand or provide signed informed consent
* Cannot provide verbal or written feedback
* Have been implanted with a pacemaker or other active medical device
* Must continuously take anticoagulants
* Uncontrolled heart or cardiovascular-related disease conditions
* Have been diagnosed with muscle atrophy and/or peripheral polyneuropathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-10; Primary Completion 2009-11 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Electrophysiological integrity of the nerves surrounded by the nerve cuffs assessed using Nerve Conduction Velocity (NCV) tests. Status Quo in physical examinations of the subject. | Throughout the study period (23 weeks)

SECONDARY OUTCOMES:
Ability to stimulate the common peroneal nerve and selectively activate ankle dorsiflexor muscles to produce symmetrical motion of the foot. Ability to sense the heel-strike and toe-lift events during walking. | From the surgical implantation to the end of the study (i.e. 20 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Dhawan, Principal Investigator — VCHA G. F. Strong Rehabilitation Centre; Michel Prud'homme, Principal Investigator — CHA- Hôpital de l'Enfant-Jésus; Ann Ashburn, Principal Investigator — University Hospital Southampton NHS Foundation Trust; Sandeep Vaishya, Principal Investigator — Max Superspeciality Hospital
Locations (4):
- Canada (2):
  - VCHA G. F. Strong Rehabilitation Centre, Vancouver, British Columbia
  - CHA- Hôpital de l'Enfant-Jésus, Québec, Quebec
- Max Superspeciality Hospital, New Delhi, New Delhi, India
- Southampton General Hospital, Southampton, Southampton, United Kingdom